CLINICAL TRIAL: NCT07305467
Title: Enhancing an Existing Prevention Strategy to Reduce Intentional Firearm Injuries Among High-risk Youth (Phase 1)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM300000392 Phase 1
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Prevention
Keywords: Firearm injury prevention; community based programs; youth advisory board

STUDY DESIGN:
Intervention Model Description: Phase I will include focus groups youth interviews (n=30) and a youth advisory board (n=15)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interviewees (Other): Interviews with youth (30 participants) to identify relevant firearm-specific risk and protective factors that will be used to develop the theory and intervention in collaboration with an advisory board of 15 youth. (Members of the YPAR are eligible to participate in both arms).
  Interventions: Other: Semi-structured focus groups
- Youth Participatory Action Research (YPAR) Advisory Board (Other): The advisory board of 15 youth. The advisory board will assist in developing the focus group protocol for Phase 1 qualitative data collection. (Members of the YPAR are eligible to participate in both arms).
  Interventions: Other: Establish an advisory board of high-risk youth; Other: Feedback and advice sessions; Other: Youth advisory board training; Other: Semi-structured focus groups

INTERVENTIONS:
Other: Establish an advisory board of high-risk youth — Fifteen high-risk youth will be recruited to establish an advisory board
  Arms: Youth Participatory Action Research (YPAR) Advisory Board
Other: Feedback and advice sessions — The youth advisory board will provide feedback and advice on the research questions, methodology, and interpretation of data through approximately fifteen, 60-minute meetings
  Arms: Youth Participatory Action Research (YPAR) Advisory Board
Other: Youth advisory board training — Youth will be trained in the social-ecological model and health behavior change theories, to better conceptualize the link between theory and intervention content, and to participate in the research process more actively.
  Arms: Youth Participatory Action Research (YPAR) Advisory Board
Other: Semi-structured focus groups — Will participate in a semi-structured focus group protocol developed in collaboration with the youth advisory board while incorporating knowledge from the empirical literature and health behavior change theories.

SUMMARY:
Over the past three decades, substantial resources have been devoted to developing youth violence prevention (YVP) programs. These programs have demonstrated positive effects on reducing aggression and related behaviors, firearm-specific risk factors were largely overlooked due to historical barriers to firearm research. This omission is concerning, as firearms are now the leading cause of injury and death among U.S. youth. Existing YVP strategies such as Emerging Leaders address general violence risk but do not directly target firearm-related risks or suicide prevention. There remains a critical gap in prevention strategies that integrate firearm-specific content while leveraging established program infrastructure.

DETAILED DESCRIPTION:
This study will utilize youth participatory action research (YPAR) to co-develop the SAFE Futures intervention. The SAFE Futures Intervention is a grounded theory of firearm-related behavior change, and it has developed the SAFE Futures single-session intervention through focus groups and youth participatory action research.

The study is designed to determine whether adding SAFE Futures to the Emerging Leaders program reduces risk factors associated with intentional firearm violence and suicide among high-risk youth. An advisory board of N=15 high-risk youth will be recruited, and data from focus groups will be analyzed using grounded theory methodology to examine attitudes, norms, personal agency, and contextual influences that promote or deter youth from engaging in risky and safe firearm behaviors (e.g., gun carrying, safe storage). The youth advisory board will use the resulting theory to develop SAFE Futures.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged approximately 13-17 years.
* Identified as at elevated risk for firearm-related injury (e.g., history of violent injury, referred by violence prevention programs).
* Able to provide assent (and parental/guardian consent if under 18).
* Sufficient proficiency in English to complete study procedures.

Exclusion Criteria:

* Significant cognitive impairment or developmental disability that would preclude comprehension of the intervention content or study procedures.
* Current psychiatric or medical instability requiring immediate treatment or hospitalization. - Non-English speaking (due to limited resources for translation of study measures and intervention materials in this pilot).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Grounded theory of firearm related change | Fifteen, 60-minute meetings (Baseline to the completion of the document)
  A document that outlines the description of the attitudes, norms, personal agency, and contextual influences that promote or deter youth from engaging in risky and safe firearm behaviors (e.g., gun carrying, safe storage), designed by the Youth Participatory Action Research (YPAR) Advisory Board during their fifteen, 60-min meetings.
SAFE Futures content | After the development of the document and through the end of the focus group development of the Intervention manual
  Intervention manual developed by the focus group interactions with the interviewees

CONTACTS AND LOCATIONS:
Overall Officials: Kelly O'Connor, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States